CLINICAL TRIAL: NCT04422782
Title: New Tools for Predicting Capillary Leak Shock During Dengue Fever
Acronym: PrediDengue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PrediDengue
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Dengue Fever; Children; Adults
Keywords: Dengue; Dengue fever; Children; Adults; French Guiana; Hypovolemic shock; Osmolarity; Hyponatremia; Hypoprotidemia; Clinical-biological score; Interstitial fluid
MeSH Terms: conditions — Dengue; Shock; Hyponatremia | interventions — Urination; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Single Arm
  Interventions: Other: For each routine sample, an additional tube will be collected to measure the osmotic pressure in the blood and urine

INTERVENTIONS:
Other: For each routine sample, an additional tube will be collected to measure the osmotic pressure in the blood and urine — Interventional research protocol involving the human person category 2 at risk and minimal constraints
  Other Names: Collection of biological samples : Aliquot of remnants of urine and blood for possible ancillary studies on prognostic factors for occurrence of shock due to capillary leakage during dengue; Systematic search for effusion done in a standardized manner with 3 ultrasound incidences: longitudinal medio axillary, longitudinal medio clavicular and transverse views of the right upper quadrant

SUMMARY:
Evaluate the prognostic value of different methods (Osmometry / clinical-biological score) compared to the occurrence of capillary leak shock during dengue fever.

DETAILED DESCRIPTION:
On the South American continent, dengue fever progressively progresses to hyperendemia with co-circulation of different serotypes. Among the complications of dengue fever, a frequent complication is the shock linked to capillary leakage which often occurs at the time of defervescence between the 3rd or 5th day of evolution of the fever. Before that, it is difficult to identify patients who are at risk for severe forms. Patients are therefore seen regularly to monitor for the development of serious forms, which causes saturation of the health system. Despite everything, with each epidemic, the investigators observe deaths of previously healthy people, which always constitutes an important trauma for the population and for the carers. Improving the understanding of the pathophysiology of capillary leakage and the tools to predict it would be significant advances in this common tropical pathology. Thus a retrospective study of longitudinal data during the dengue 2 epidemic of 2013 made it possible to generate precise hypotheses as to the pathophysiology of the shock linked to capillary leakage. Hypoprotidemia and hyponatremia having a strong statistical association with the subsequent occurrence of shock, the hypothesis is of a progressive disturbance of the plasma osmolarity resulting in water leaks towards the interstitial sector.

These preliminary data also made it possible to develop a predictive score which must now be validated over time.

Research involving the human person, monocentric, prospective, validation

Interventional research protocol involving the human person category 2 at risk and minimal constraints

ELIGIBILITY:
Inclusion Criteria:

* Age> = 5 years
* Patient / parent consent
* Exclude other pathology with capillary circulation problem (septic shock, anaphylaxis) All suspected dengue fever requiring hospitalization will be included, final inclusion being after biological confirmation (AgNS1, RT-PCR, serology).

Exclusion Criteria:

* Age <5 years
* Refusal to participate
* Unsigned consent
* Coinfection by another agent
* Patient under guardianship or curatorship.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2022-05-14 (Estimated); Study Completion 2023-05-14 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a shock | 2 years
  The primary outcome measure will be the occurrence of a shock defined by systolic blood pressure <90 mm Hg in adults and <80 mm Hg in children.

SECONDARY OUTCOMES:
Predictive value of plasma hypo-osmolarity | 2 years
  Evaluate the predictive value of plasma hypo-osmolarity in the occurrence of shock during dengue
Validation of the clinical-biological prognostic score | 2 years
  Prospectively validate the clinical-biological prognostic score (2013 shock score) and, if possible, improve it
Relationship between the measurements obtained by osmolarity and capillary leakage | 2 years
  Study the relationship between the measurements obtained by osmolarity and capillary leakage measured by pleural effusion
Evaluation of the sensitivity / specificity and predictive values of osmolarity and capillary leakage | 2 years
  Evaluation of the sensitivity / specificity and predictive values of these measures in relation to the ultrasound objectification of a pleural effusion
How long before the shock these measures (osmolarity, score) allow to predict an unfavorable evolution | 2 years
  Specify how long before the shock these measures (osmolarity, score) allow to predict an unfavorable evolution
Association between the factor "Presence of sickle cell disease" and "occurrence of severe dengue" | 2 years
  Study the association between the factor "Presence of sickle cell disease" and "occurrence of severe dengue"

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, MD, PhD, Study Director — Centre Hospitalier de Cayenne
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana, France

REFERENCES:
- [Background] Djossou F, Vesin G, Elenga N, Demar M, Epelboin L, Walter G, Abboud P, Le-Guen T, Rousset D, Moreau B, Mahamat A, Malvy D, Nacher M. A predictive score for hypotension in patients with confirmed dengue fever in Cayenne Hospital, French Guiana. Trans R Soc Trop Med Hyg. 2016 Dec 1;110(12):705-713. doi: 10.1093/trstmh/trx004. PMID 28938048